CLINICAL TRIAL: NCT02571842
Title: A Randomized, Prospective, Open-Label Study of Rituximab in the Treatment of Recurrent IgA Nephropathy With Active Endocapillary Proliferation Pathology
Brief Title: Rituximab in Recurrent IgA Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wiwat Chancharoenthana, Dr., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WWC-006
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Recurrent IgA Nephropathy
Keywords: Recurrent IgA nephropathy; Rituximab
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Rituximab; Adrenal Cortex Hormones; Enalapril; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Drug: Rituximab
  •Rituximab 375 mg/m2 on treatment month 1, 2, 3, 4
  Other Name: Mabthera
  Interventions: Drug: Intravenous Rituximab
- ACEI/ARB plus corticosteroids (Active Comparator): Drug: ACEI/ARB
  * An ACEI and /or ARBs will be used to achieve proteinuria reduction and a blood pressure goal of <130/80 mmHg. Patients not attaining the target blood pressure with an ACEI or ARB alone should be treated with the combination of ACEI + ARB
  * Corticosteroids will be used as prednisolone 0.5 mg/kg/day with gradually taper off in 6-8 weeks to 5mg/day daily
  Other Name: Enalapril, Lorsartan, Prednisolone
  Interventions: Drug: ACEI/ARB and corticosteroids

INTERVENTIONS:
Drug: Intravenous Rituximab — - 375 mg/m2 rituximab be prescribed 4 consecutive monthly
  Other Names: Mabthera
  Arms: Rituximab
Drug: ACEI/ARB and corticosteroids — * ACEI or ARB will be prescribed as high as tolerable dose.
  * Prednisolone will be prescribed starting as 0.5 mg/kg/day then taper off to 5 mg/day within 6-8 weeks
  Other Names: "Enalapril", "Lorsartan", "Prednisolone
  Arms: ACEI/ARB plus corticosteroids

SUMMARY:
Currently, the treatment options of recurrent IgA nephropathy (IgAN) are conflicting and largely based on expert opinions. Consequently, the recent KDIGO clinical practice guideline for the care of kidney transplant recipients has concluded that there are no definite strategies for prevention and treatment. However, recurrent IgAN in the transplanted kidney is common and may contribute to graft loss, in particular, if cresentic formation, extra- or endocapillary proliferation were presented in kidney pathology. Herein, the investigators assume that rituximab, anti-CD20 Ab agent, can reduce circulating IgA with subsequently decrease rate of polymeric forms of IgA deposition in glomerular capillaries. Therefore, the investigators speculate that rituximab may have potential effect to reduce circulating polymeric forms of IgA and slow progression of recurrent IgAN.

DETAILED DESCRIPTION:
Hypothesis: In kidney transplant recipients with active endocapillary proliferation pathology of recurrent IgAN, an intravenous infusion of 375mg/m2 of rituximab on 4 consecutive monthly dose is superior to conventional therapy in reducing 24-hour proteinuria, and slowing progression of recurrent IgAN.

ELIGIBILITY:
Inclusion Criteria:

* Any kidney transplant recipients between the age of 18 and 70 years of age and able to give informed consent
* GFR by 24h Creatinine Clearance (CrCl) >30 ml/min/1.73m²
* Biopsy proven recurrent IgA nephropathy with endocapillary proliferation pattern

Exclusion Criteria:

* Clinical and histologic evidence of IgA combination with other forms of glomerulonephritis
* Clinical evidence of cirrhosis, chronic active liver disease or known infection with hepatitis B, C or HIV
* 24h CrCl <30 ml/min/1.73m² at the time of screening
* Active systemic infection or history of serious infection within one month of entry
* Positive pregnancy test or breast feeding at time of study entry
* Patients receiving >6 months therapy with oral prednisone >5mg/day or glucocorticoid equivalent
* Live vaccine within 28 days of study enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Remission rate | 12 months
  Percentage of patients in each group achieving complete or partial response determined by proteinuria and 24-hour creatinine clearance
Incidence of all adverse events | 12 months
  The incidence of adverse events such as serious infection, allergy, fever, headache, etc.

SECONDARY OUTCOMES:
Change in allograft pathology following treatment | 12 months
  The difference of active and chronic score report by BANFF score, HAAS, Oxford criteria between pre-treatment and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wiwat Chancharoenthana, M.D., Ph.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Bangkok, Thailand